CLINICAL TRIAL: NCT04079400
Title: Microbiome in Patients With Pulmonary Tuberculosis, Non-tuberculous Mycobacterial Pulmonary Diseases (NTM-PD), Lung Cancer and Hemoptysis
Brief Title: Microbiome in Pulmonary Tuberculosis, Non-tuberculous Mycobacterial Pulmonary Diseases, Lung Cancer and Hemoptysis
Status: Completed | Type: Observational
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Sangmin Lee, MD, Associate professor, Gachon University Gil Medical Center
Other Study IDs: 2016-5205
Record Dates: First submitted 2019-09-03; First posted 2019-09-06 (Actual); Last update posted 2019-09-06 (Actual); Status verified 2019-09

CONDITIONS: Tuberculosis, Pulmonary; Non-Tuberculous Mycobacterial Pneumonia; Lung Cancer; Hemoptysis
MeSH Terms: conditions — Tuberculosis, Pulmonary; Lung Neoplasms; Hemoptysis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Lower respiratory specimens acquired by bronchial brushing and washing for 16S rRNA sequencing
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- Tb group: Subjects who underwent bronchoscopy for suspicious endobronchial pulmonary tuberculosis (Tb) observed on chest computed tomography
- NTM-PD group: Subjects who underwent bronchoscopy for suspicious non-tuberculous mycobacterial pulmonary disease (NTM-PD) observed on chest computed tomography
- LC group: Subjects who underwent bronchoscopy for suspicious endobronchial lung cancer (LC) observed on chest computed tomography
- HM group: Subjects who underwent bronchoscopy for hemoptysis
- Control group: Subjects who underwent bronchoscopy to rule out endobronchial lesion observed on chest computed tomography. Endbronchial lesion should not be typical for any category of respiratory diseases including tuberculosis, NTM-TB and lung cancer.

SUMMARY:
Microbiome in lower respiratory diseases is not sufficiently known yet. The objective of this study is to investigate microbiome in patients who present with hemoptysis, and those with pulmonary tuberculosis, non-tuberculous mycobacterial pulmonary disease (NTM-PD), and lung cancer, analyzing respiratory specimen acquired by bronchoscopic approach.

DETAILED DESCRIPTION:
Subjects who were going to undergo bronchoscopy for hemoptysis or suspected lower respiratory diseases including endobronchial tuberculosis (Tb), NTM-PD, or endobronchial lung cancer (LC) were enrolled after informed consents.

Subjects who were supposed to receive bronchoscopy to rule out endobronchial lesions were also enrolled as control group (ctrl) after informed consents. In those control group, endobronchial tuberculosis, malignancy or other certain respiratory diseases was not clearly suspected.

Before acquiring respiratory specimens, bronchoscopic channels were washed to acquire negative control in all cases of groups.

In Tb group and LC group, specimens of normal bronchial mucosa near suspicious endobronchial lesion were obtained with protected brush (PB), then specimens of abnormal bronchial mucosa in suspicious endobronchial lesion with PB. After acquiring respiratory specimens of PB, bronchial washing was done in suspicious endobronchial lesion.

In NTM-PD group, specimens of bronchial mucosa in bronchus of suspicious NTM-PD with PB. After acquiring respiratory specimens of PB, bronchial washing was done in bronchus of suspicious NTM-PD.

In hemoptysis group, bronchial washing was done in bronchus of ongoing bleeding.

In control group, specimens of bronchial mucosa in predetermined random bronchus (not bronchus with suspicious endobronchial lesion) with PB. After acquiring respiratory specimens of PB, bronchial washing was done in the same bronchus.

Microbiome in lower respiratory species was analyzed using 16S rRNA sequencing.

ELIGIBILITY:
Inclusion Criteria:

* Patients who underwent bronchoscopy for hemoptysis, OR
* Patients who underwent bronchoscopy for suspicious endobronchial pulmonary tuberculosis observed on chest computed tomography, OR
* Patients who underwent bronchoscopy for suspicious non-tuberculous mycobacterial pulmonary disease (NTM-PD) observed on chest computed tomography, OR
* Patients who underwent bronchoscopy for suspicious endobronchial lung cancer observed on chest computed tomography, OR
* Patients who underwent bronchoscopy to rule out endobronchial lesion which did not seem to be typical for any criteria of pulmonary diseases including tuberculosis, NTM-PD or lung cancer on chest computed tomography

Exclusion Criteria:

* Other malignancy, infection or serious diseases of neural, cardiovascular, renal, hepatobiliary, gastrointestinal, hemotologic or respiratory system
* Use of any antibiotic within a month
* Vulnerable volunteer
* Subject's rejection

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. HM group
     * Patients who underwent bronchoscopy for hemoptysis
  2. Tb group
     * Patients who underwent bronchoscopy for suspicious endobronchial pulmonary tuberculosis
  3. NTM-PD group
     * Patients who underwent bronchoscopy for suspicious non-tuberculous mycobacterial pulmonary disease (NTM-PD)
  4. LC group
     * Patients who underwent bronchoscopy for suspicious endobronchial lung cancer
  5. Control group
     * Patients who underwent bronchoscopy to rule out endobronchial lesion which did not seem to be typical for any criteria of pulmonary diseases including tuberculosis, NTM-PD or lung cancer
Sampling Method: Non-Probability Sample
Enrollment: 43 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2019-04-11 (Actual)

PRIMARY OUTCOMES:
16S rRNA sequencing | 0 day (the day of study enrollment)
  The V1 to V3 regions of the 16S rRNA in respiratory specimens were analyzed for identification of microbiomes.

CONTACTS AND LOCATIONS:
Overall Officials: Sang Min Lee, MD, PhD, Principal Investigator — Gachon Univ. Gil Medical Center

IPD SHARING:
Plan to Share IPD: No
Technically, results of 16S rRNA sequencing can hardly be shared. Study protocol, SAP, ICF, CSR were written in Korean, so they can not be shared either.

REFERENCES:
- [Background] Caverly LJ, Carmody LA, Haig SJ, Kotlarz N, Kalikin LM, Raskin L, LiPuma JJ. Culture-Independent Identification of Nontuberculous Mycobacteria in Cystic Fibrosis Respiratory Samples. PLoS One. 2016 Apr 19;11(4):e0153876. doi: 10.1371/journal.pone.0153876. eCollection 2016. PMID 27093603
- [Background] Green H, Jones AM. The microbiome and emerging pathogens in cystic fibrosis and non-cystic fibrosis bronchiectasis. Semin Respir Crit Care Med. 2015 Apr;36(2):225-35. doi: 10.1055/s-0035-1546752. Epub 2015 Mar 31. PMID 25826590
- [Background] Tunney MM, Einarsson GG, Wei L, Drain M, Klem ER, Cardwell C, Ennis M, Boucher RC, Wolfgang MC, Elborn JS. Lung microbiota and bacterial abundance in patients with bronchiectasis when clinically stable and during exacerbation. Am J Respir Crit Care Med. 2013 May 15;187(10):1118-26. doi: 10.1164/rccm.201210-1937OC. PMID 23348972
- [Background] Yu G, Gail MH, Consonni D, Carugno M, Humphrys M, Pesatori AC, Caporaso NE, Goedert JJ, Ravel J, Landi MT. Characterizing human lung tissue microbiota and its relationship to epidemiological and clinical features. Genome Biol. 2016 Jul 28;17(1):163. doi: 10.1186/s13059-016-1021-1. PMID 27468850
- [Result] Philley JV, Kannan A, Olusola P, McGaha P, Singh KP, Samten B, Griffith DE, Dasgupta S. Microbiome Diversity in Sputum of Nontuberculous Mycobacteria Infected Women with a History of Breast Cancer. Cell Physiol Biochem. 2019;52(2):263-279. doi: 10.33594/000000020. Epub 2019 Feb 28. PMID 30816674
- [Result] Cheung MK, Lam WY, Fung WY, Law PT, Au CH, Nong W, Kam KM, Kwan HS, Tsui SK. Sputum microbiota in tuberculosis as revealed by 16S rRNA pyrosequencing. PLoS One. 2013;8(1):e54574. doi: 10.1371/journal.pone.0054574. Epub 2013 Jan 24. PMID 23365674
- [Result] Adami AJ, Cervantes JL. The microbiome at the pulmonary alveolar niche and its role in Mycobacterium tuberculosis infection. Tuberculosis (Edinb). 2015 Dec;95(6):651-658. doi: 10.1016/j.tube.2015.07.004. Epub 2015 Jul 30. PMID 26455529
- [Result] Lee SH, Sung JY, Yong D, Chun J, Kim SY, Song JH, Chung KS, Kim EY, Jung JY, Kang YA, Kim YS, Kim SK, Chang J, Park MS. Characterization of microbiome in bronchoalveolar lavage fluid of patients with lung cancer comparing with benign mass like lesions. Lung Cancer. 2016 Dec;102:89-95. doi: 10.1016/j.lungcan.2016.10.016. Epub 2016 Oct 31. PMID 27987594
- [Result] Yan X, Yang M, Liu J, Gao R, Hu J, Li J, Zhang L, Shi Y, Guo H, Cheng J, Razi M, Pang S, Yu X, Hu S. Discovery and validation of potential bacterial biomarkers for lung cancer. Am J Cancer Res. 2015 Sep 15;5(10):3111-22. eCollection 2015. PMID 26693063
- [Result] Vogtmann E, Goedert JJ. Epidemiologic studies of the human microbiome and cancer. Br J Cancer. 2016 Feb 2;114(3):237-42. doi: 10.1038/bjc.2015.465. Epub 2016 Jan 5. PMID 26730578
- [Result] Hosgood HD 3rd, Sapkota AR, Rothman N, Rohan T, Hu W, Xu J, Vermeulen R, He X, White JR, Wu G, Wei F, Mongodin EF, Lan Q. The potential role of lung microbiota in lung cancer attributed to household coal burning exposures. Environ Mol Mutagen. 2014 Oct;55(8):643-51. doi: 10.1002/em.21878. Epub 2014 Jun 3. PMID 24895247
- [Result] Liu HX, Tao LL, Zhang J, Zhu YG, Zheng Y, Liu D, Zhou M, Ke H, Shi MM, Qu JM. Difference of lower airway microbiome in bilateral protected specimen brush between lung cancer patients with unilateral lobar masses and control subjects. Int J Cancer. 2018 Feb 15;142(4):769-778. doi: 10.1002/ijc.31098. Epub 2017 Nov 8. PMID 29023689